CLINICAL TRIAL: NCT07362706
Title: An Exploratory Study on the Impact of Prolonged Postoperative Endotracheal Extubation Time on Postoperative Complications in Gastric Cancer Patients With Severe Obstructive Sleep Apnea
Brief Title: Prolonged Extubation in Gastric Cancer With OSA
Acronym: Gastric Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202110-034-2
Record Dates: First submitted 2025-08-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea; Gastric Cancer (GC)
Keywords: Radical gastrectomy; Severe obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Prolonging the duration of postoperative endotracheal intubation before extubation. — The patients were divided into two groups, the extended tracheal intubationremoval time group (24-48h)and the non-extended tracheal intubation removal time group, and the incidenceof surgery-related complications and non-surgical-related complications in the two groups werecompared.

SUMMARY:
This study aims to investigate the effect of prolonged tracheal intubation removal on the incidenceof postoperative complications in patients with gastric cancer complicated with severe obstructive sleepapnea.

DETAILED DESCRIPTION:
This study retrospectively included patients who underwent radical gastrectomycombined with severe obstructive sleep apnea at Qilu Hospital . Accordingto the assessment of anesthesiologists, whether the anesthetic drugs of the patients were adequatelymetabolized during the operation. The patients were divided into two groups, the extended tracheal intubationremoval time group (24-48h)and the non-extended tracheal intubation removal time group, and the incidenceof surgery-related complications and non-surgical-related complications in the two groups werecompared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients preoperatively diagnosed with resectable gastric cancer
2. Patients without distant organ metastasis
3. Patients with preoperative Overnight Cardiorespiratory Sleep Testing (OCST) or Polysomnography (PSG) results showing Apnea-Hypopnea Index (AHI) >30 events/hour and SaO₂ <80%
4. Patients with cardiopulmonary function deemed suitable for surgery
5. Patients aged 18-85 years
6. Patients who voluntarily joined this study and provided written informed consent

Exclusion Criteria:

1. Patients with a history of or concurrent other malignant tumors
2. Patients who underwent palliative resection
3. Subjects who experienced acute cardiovascular or cerebrovascular events (e.g., acute cerebral infarction, acute coronary syndrome) within the past 3 months, or whose cardiovascular clinical symptoms/diseases are not well-controlled
4. Patients with a history of psychotropic drug abuse that cannot be abstained, or those with psychiatric disorders
5. Patients with concomitant diseases that, in the investigator's judgment, seriously endanger the patient's safety or affect the completion of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer complicated with severe sleep apnea
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 48-72 hour
  The incidence of postoperative complications in patients with gastric cancer complicated with severe obstructive sleepapnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

DOCUMENTS (1):
  • Study Protocol (2026-01-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT07362706/Prot_000.pdf